CLINICAL TRIAL: NCT03705260
Title: Achieving Improved Control of Blood Glucose Among Type 2 Diabetes Patients Through Continuous Glucose Monitoring & Care Coordinator Mediated Gains in Patient Self-Management Sophistication
Brief Title: Quality Initiative to Improve Glucose Control in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Twine Clinical Consulting (Unknown)
Responsible Party: Principal Investigator, Caroline Richardson, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00147295
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Comparator- High Risk (Active Comparator): A high risk sub group of those assigned to the comparator arm will be identified by their most recent A1C > 8. Patients in this group will receive usual care from their Primary Care Physician and dietitian.
  Interventions: Other: Usual Care
- Comparator- Well Controlled (Active Comparator): The low risk sub group from the comparator arm (A1C < 8) and those who are unlikely to benefit from an intensive behavioral intervention will get usual care by their Primary Care Physician and their dietitian.
  Interventions: Other: Usual Care
- Enhanced Care- High Risk (Experimental): A high risk sub group of those assigned to the enhanced care arm will be identified by their most recent A1C > 8. Patients in this group will receive the intensive behavioral intervention which will incorporate lower carbohydrate diet, diet coaching, and more intensive glucose monitoring.
  Interventions: Behavioral: Intensive Behavioral Intervention
- Enhanced Care- Well Controlled. (Experimental): The low risk sub group from the enhanced care arm (A1C < 8) and those who are unlikely to benefit from an intensive behavioral intervention will get usual care by their PCP and their dietitian. If they are found to be poorly controlled through monthly screening for risk, they may have the opportunity to move into the Enhanced Care High Risk group.
  Interventions: Other: Usual Care; Other: Monthly Screening for Risk

INTERVENTIONS:
Other: Usual Care — Usual care from Primary Care Physician and dietitian.
  Arms: Comparator- High Risk; Comparator- Well Controlled; Enhanced Care- Well Controlled.
Behavioral: Intensive Behavioral Intervention — The intensive behavioral intervention which will incorporate lower carbohydrate diet, diet coaching, and more intensive glucose monitoring.
  Arms: Enhanced Care- High Risk
Other: Monthly Screening for Risk — Monthly screening of HbA1C to identify patents who have become poorly controlled in the interval.
  Arms: Enhanced Care- Well Controlled.

SUMMARY:
The goal of the Twine / University of Michigan Diabetes Quality Improvement Initiative is to improve diabetes care quality using real time feedback with continuous glucose monitoring (CGM) and dietary coaching for lower carbohydrate consumption in a high-risk sub-cohort of outpatients with type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Michigan Medicine patient treated by a physician in the Family Medicine Department at the Chelsea Health Center
* Diagnosis of T2D as recorded in the patient's problem list or as documented by medication list and lab results
* HbA1C >8 for the high-risk sub-cohort

Exclusion Criteria:

* Individuals for whom tight control (ie A1C < 8) is not safe or recommended, including but not limited to older frail individuals at high-risk of hypoglycemia and falls or those with a life expectancy of less than 6 months due to a comorbid condition
* Individuals with cognitive or psychological diagnoses that might make CGM or low carbohydrate dieting risky, such as patients with eating disorders, uncontrolled psychotic - mental illness or those patients with dementia
* Women who are pregnant or breast feeding
* Individuals who had previous bariatric surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | 1 year
  Hemoglobin A1C

SECONDARY OUTCOMES:
Weight Change | baseline to 1 year
  Difference in patient's weight measured in pounds.
Change in diabetes medication requirements | baseline to 1 year
  Change in average daily doses of diabetes medications
Change in percentage of time glucose is out of range | baseline to 1 year
  Change in percentage of time glucose is out of range (70 mg/dl-140 mg/dl) on CGM.
Blood Pressure | 1 year
  Blood Pressure
Change in rate of Micro-vascular complications | Baseline to 1 Year
  Change in rate of micro-vascular complications. (The micro-vascular complications assessed will be retinopathy, neuropathy, nephropathy)
Change in rate of symptomatic hypoglycemia requiring medical intervention | Baseline to 1 year
  Change in rate of symptomatic hypoglycemia requiring medical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Richardson, M.D., Principal Investigator — University of Michigan
Locations (1):
- Chelsea Health Center, Chelsea, Michigan, United States

IPD SHARING:
Plan to Share IPD: No